CLINICAL TRIAL: NCT02647957
Title: Indicators for Quality Assessment of Hospitalized Ischemic Stroke Patients. A Study of the Efficacy of the Code Stroke in Spain
Brief Title: A Study of the Efficacy of the Code Stroke in Spain
Acronym: QICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital Serranía de Ronda (Unknown); Hospital of Navarra (Other); Hospital Virgen de la Concha (Unknown); Hospital of Jaen (Other); Hospital General San Jorge (Unknown)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 489/2015
Record Dates: First submitted 2015-12-26; First posted 2016-01-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Stroke, Acute
Keywords: acute ischemic stroke; quality
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Hospital using Code Stroke
  Interventions: Procedure: Code Stroke
- Group B (No Intervention): Hospital not using Code Stroke

INTERVENTIONS:
Procedure: Code Stroke — Apply a protocol called Code Stroke that involves the entire care chain from emergency teams outpatient specialists of Neurology, Internal Medicine, Radiology or Intensitivos Care, among other hospital areas.
  Arms: Group A

SUMMARY:
Code Stroke is a system for the rapid identification, pre-notification and transport of acute ischemic stroke patients. The objective of this study was to define quality indicators and to compare treatment outcomes in hospitals where Code Stroke has been implemented and hospitals without the use of Code Stroke (control patients).

DETAILED DESCRIPTION:
In a first step qualitative technique has been conducted to define treatment quality indicators of acute ischemic stroke patients. In a second step a prospective study is conducted to collect data of 240 inpatients from two groups of hospitals. Two hospitals applying Code Stroke (N= 120) and four hospitals non-applying Code Stroke procedure (N=120). A consecutive sampling method will be conducted. Inclusion criteria: acute ischemic stroke patients treated in the hospitals during the field study. The referral to the hospital could be from primary care, Emergency Unit of other hospital. Patients will enroll after inform consent.

A Singer-blind- research method will applied. Quality indicators defined in the first phase will be applied and comparisons will be realized using ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke in-patients

Exclusion Criteria:

* Patients who refuse participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recovery rate of the Intravenous trombolysis treatment | 1 month
  Number of patients showing an adequate recovery after Intravenous trombolysis treatment as assessed by the criteria of the Quality Indicator Board of the German Stroke Registers Study Group and the National Sentinel Audit of Stroke.

SECONDARY OUTCOMES:
Patient satisfaction | 1 month
  Patient Satisfaction Scale
Patient engage | 1 month
  Health literacy Scale
response capacity | 1 day
  Response time for the initial evaluation and treatment
Treatment adequacy: Intravenous trombolysis treatment | 1 month
  Intravenous trombolysis treatment applied in eligible ischemic stroke patients
Patient safety. Complications in the recombinant tissue plasminogen activator treatment after tromobysis | 1 month
  Recombinant tissue plasminogen activator complication rates
Mortality rates of the Intravenous trombolysis treatment | 1 month
  Mortality rates of the Intravenous trombolysis treatment when applied in eligible ischemic stroke patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez Sabin J, Molina C, Abilleira S, Montaner J, Garcia F, Alijotas J. ["Stroke code". Shortening the delay in reperfusion treatment of acute ischemic stroke]. Med Clin (Barc). 1999 Oct 23;113(13):481-3. Spanish. PMID 10604170